CLINICAL TRIAL: NCT02294526
Title: PILCHARDUS STUDY: A Sardine Diet Intervention Study to Assess Benefits to the Metabolic Profile in Type 2 Diabetes Mellitus Patients
Brief Title: A Sardine Diet Intervention Study to Assess Benefits to the Metabolic Profile in Type 2 Diabetes Mellitus Patients
Acronym: PILCHARDUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spanish Biomedical Research Centre in Diabetes and Associated Metabolic Disorders (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIBERDEM-PILCHARDUS
Record Dates: First submitted 2014-10-31; First posted 2014-11-19 (Estimated); Last update posted 2015-01-29 (Estimated); Status verified 2014-11

CONDITIONS: Type 2 Diabetes
Keywords: Diet; Sardine; Type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sardine diet (Experimental): Subjects follow general dietary recommendations for diabetes including a fixed amount of sardine in daily meals (100g per day, 5 days a week) as part of their usual diet.
  Interventions: Other: Sardine diet
- Control diet (No Intervention): Subjects only follow general dietary recommendations for diabetes.

INTERVENTIONS:
Other: Sardine diet — Diet rich in sardine: 100g/day of sardine 5 times a week
  Arms: Sardine diet

SUMMARY:
Work hypothesis

A diet rich in sardine will improve the metabolic control in type 2 diabetes patients.

ELIGIBILITY:
Inclusion Criteria:

* Age > 40 years and < 85
* BMI ≥ 25 and < 35
* Patients diagnosed with type 2 diabetes at onset or treated only by diet
* HbA1c between 6.0 and 8.0% (based on the last measured and documented laboratory measurement of the previous 3 months)
* Usual consumption ≤ 3 fish per week

Exclusion Criteria:

* T2D treated with antidiabetic oral drugs and/or insulin
* Current or previous (within 3 months) intake of omega 3 suplements
* Known allergy or intolerance to fish or fish protein
* Diagnosis of active neoplasic disease
* Suffering from an acute illness which requires a recovery period higher than one week
* Currently chronic treatment with oral steroids or nonesteroidal anti-inflammatory for more than 5 days, at least 1 month before randomization
* Pregnant or breast-feeding patients
* Serious acute vascular events (cardiac or cerebral) diagnosed previous 2 months before the randomization
* Current or previous (within 6 months) participation in another study
* Chronic renal insufficiency (creatinine >1,5 mg/dl)
* Any conditions that the investigator considers may render the patient unable to complete the study

During the interventional study, based on current standards of T2D care, doctors will introduce anti-diabetic oral drugs or insulin into the patient's treatment, where they consider it to be necessary.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2012-11; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline in glycated hemoglobin (HbA1c) at 6 months | Baseline and 6 months
Change from baseline in fasting glucose at 6 months | Baseline and 6 months
Change from baseline in fasting insulin at 6 months | Baseline and 6 months

SECONDARY OUTCOMES:
Change from baseline in adiponectin at 6 months | Baseline and 6 months
Change from baseline in leptin at 6 months | Baseline and 6 months
Change from baseline in ultra sensitive C-reactive protein (us-CRP) at 6 months | Baseline and 6 months
Change from baseline in interleukin-6 (IL-6) at 6 months | Baseline and 6 months
Change from baseline in interleukin-8 (IL-8) at 6 months | Baseline and 6 months
Change from baseline in interleukin-10 (IL-10) at 6 months | Baseline and 6 months
Change from baseline in tumor necrosis factor alpha (TNFα) at 6 months | Baseline and 6 months
Change from baseline in erytrocite membrane fatty acid composition (EMFA) at 6 months | Baseline and 6 months
Change from baseline in specific bacterial groups of gut microbiota at 6 months | Baseline and 6 months
Change from baseline in total cholesterol at 6 months | Baseline and 6 months
Change from baseline in LDL cholesterol at 6 months | Baseline and 6 months
Change from baseline in HDL cholesterol at 6 months | Baseline and 6 months
Change from baseline in triglycerides at 6 months | Baseline and 6 months
Change from baseline in blood pressure at 6 months | Baseline and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Ramon Gomis, Professor, Principal Investigator — CIBERDEM - IDIBAPS (Institut d'Investigacions Biomèdiques August Pi i Sunyer) - Hospital Clínic of Barcelona

REFERENCES:
- [Derived] Balfego M, Canivell S, Hanzu FA, Sala-Vila A, Martinez-Medina M, Murillo S, Mur T, Ruano EG, Linares F, Porras N, Valladares S, Fontalba M, Roura E, Novials A, Hernandez C, Aranda G, Siso-Almirall A, Rojo-Martinez G, Simo R, Gomis R. Effects of sardine-enriched diet on metabolic control, inflammation and gut microbiota in drug-naive patients with type 2 diabetes: a pilot randomized trial. Lipids Health Dis. 2016 Apr 18;15:78. doi: 10.1186/s12944-016-0245-0. PMID 27090218